CLINICAL TRIAL: NCT02870829
Title: Treatment to Reduce Vascular Calcification in Hemodialysis Patients Using Vitamin K (Trevasc-HDK): A Study Protocol for a Randomized Controlled Trial
Brief Title: Treatment to Reduce Vascular Calcification in Hemodialysis Patients Using Vitamin K
Acronym: TReVasc-HDK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); Nattopharma ASA (Industry)
Responsible Party: Principal Investigator, Sabrina Haroon Wong Peixin, Consultant Nephrologist, University Medicine Cluster, National University Health System, Singapore
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHG DSRB Ref: 2015/01000
Record Dates: First submitted 2016-08-14; First posted 2016-08-17 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Vascular Calcification; Systemic and Arterial Stiffness; Complication of Hemodialysis; Deficiency of Vitamin K2
MeSH Terms: conditions — Vascular Calcification | interventions — menaquinone 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin K2 (Experimental): Vitamin K comes in various isoforms and we have elected to use the K2 isoform - menaquinone-7. We have chosen a dose of 360mcg 3x/week as previous studies using menaquinone-7 demonstrated an increasing dose efficacy relationship up to this strength. Vitamin K2 is manufactured by Nattopharma
  Interventions: Drug: menaquinone-7
- Standard Therapy (No Intervention): Subjects randomised to standard therapy will continue to receive dialysis and chronic kidney disease-metabolic bone disease (CKD-MBD) management in accordance to current best practise guidelines

INTERVENTIONS:
Drug: menaquinone-7 — Oral supplement given post dialysis 3x/week
  Arms: Vitamin K2

SUMMARY:
The proposed study will seek to evaluate the prevalence and the progression of vascular calcification in a cohort of maintenance hemodialysis patients in Asian population. It will also evaluate the efficacy of vitamin K 2 supplementation in reducing the progression of vascular calcification in this group of patients.

This will be a single-center randomized, prospective and open-label interventional clinical trial of end stage renal failure patients on hemodialysis.Primary outcome will be absolute difference in coronary artery calcium (CAC) score at 18-month between control and intervention arms. Secondary outcomes will be to compare absolute difference in aortic valve calcification, percentage of patients with regression of coronary artery calcification of at least 10%, absolute difference in aortic and systemic arterial stiffness, mortality from any cause and major adverse cardiovascular events (MACE) over the same period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 years and less than 80 years
2. At least 12 months on Hemodialysis
3. Coronary artery calcium score of ≥ 30 in the baseline Multislice Computed Tomography
4. Able to give informed consent
5. Life expectancy of at least18 months

Exclusion Criteria:

1. History of thrombosis in the last 6 months except vascular access thrombosis
2. Need for vitamin K antagonists therapy at baseline or in the 3 months prior to baseline
3. Presence of significant gut disease (inflammatory bowel disease, short-bowel syndrome)
4. Liver dysfunction
5. Alcohol or drug abuse
6. Presence of coronary stent or have undergone coronary artery bypass grafting
7. Women who are pregnant or breast feeding,
8. Those who are fearful of confined space and cannot lie still for Multislice Computed Tomography
9. Lack of safe contraceptive measures.
10. Those who had parathyroid surgery done.
11. Those with parathyroid hormone (PTH) > 150 pmol/l
12. Patient taking multivitamins containing vitamin K
13. Patient allergic to soy based products

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Absolute difference in coronary artery calcium score at 18-month between control and intervention arms | 18 months
  Comparison made using the t-test following log transformation. Adjustment for baseline CAC scores made via the analysis of covariance.

SECONDARY OUTCOMES:
Absolute difference in AVC score at 18-months | 18 months
  Comparison made using the t-test following log transformation. Adjustment for baseline AVC scores made via the analysis of covariance.
Percentage of patients with regression of CAC of ≥ 10% over 18-month | 18 months
Absolute difference in cfPWV and AI at 18-months | 18 months
Mortality from any cause within the study period | 18 months
MACE defined as non-fatal myocardial infarction, heart failure, acute coronary syndrome, need for coronary revascularization, non-fatal stroke, significant peripheral vascular disease | 18 months
Difference in plasma levels of dp-ucMGP at 18 months | 18 months
Vascular access events, including clotting requiring insertion of a new dialysis catheter, declotting or exchange of an existing catheter, and vascular intervention during the study period | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Wong Peixin Haroon, MD MRCP FAMS, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared with collaborators

REFERENCES:
- [Derived] Haroon SW, Tai BC, Ling LH, Teo L, Davenport A, Schurgers L, Teo BW, Khatri P, Ong CC, Low S, Yeo XE, Tan JN, Subramanian S, Chua HR, Tan SY, Wong WK, Lau TW. Treatment to reduce vascular calcification in hemodialysis patients using vitamin K (Trevasc-HDK): A study protocol for a randomized controlled trial. Medicine (Baltimore). 2020 Sep 4;99(36):e21906. doi: 10.1097/MD.0000000000021906. PMID 32899022